CLINICAL TRIAL: NCT02409238
Title: Insulin Resistance and Mild Cognitive Impairment (MCI) in Older Chinese Adults With Pre-Diabetes and Diabetes: Cognitive Effects of Lifestyle Intervention and Metformin Treatment in a Randomized Controlled Trial
Brief Title: Insulin Resistance and Mild Cognitive Impairment (IRMCI) Study
Acronym: IRMCI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 1. Limits of grant funding reached
  2. A/Prof Ng Tze Pin (P.I. & holder of NMRC Grant (CIRG12may033) funding this study) retired in Aug 2022.
  3. Resignations of staff and collaborators especially over the 1st 2 years of the COVID-19 pandemic
Sponsor: SingHealth Polyclinics (Other)
Collaborators: National University of Singapore (Other); Singapore General Hospital (Other); Changi General Hospital (Other); National University Hospital, Singapore (Other); Singapore Clinical Research Institute (Other); Agency for Science, Technology and Research (Other); Khoo Teck Puat Hospital (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Andrew Wee Kien Han, Family Physician- SITE Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCI-LM 3
Record Dates: First submitted 2015-03-26; First posted 2015-04-06 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment; Insulin Resistance; Diabetes Mellitus, Type 2
Keywords: Mild Cognitive Impairment; Insulin Resistance; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Cognitive Dysfunction; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Intervention and Metformin (Experimental): Intensive lifestyle interventions at Lifestyle Intervention Centres and Metformin (if Diabetic)
  Interventions: Drug: Metformin; Behavioral: Intensive Lifestyle Intervention
- Standard Level of Care (Active Comparator): Standard lifestyle recommendations for the Control groups
  Interventions: Behavioral: Standard LIfestyle Recommendation

INTERVENTIONS:
Drug: Metformin — Metformin dosage schedule: 250 mg thrice a day titrated from 250 mg once a day. Patients will first be started on Metformin 250 mg once a day with meals, and the dose increased to 250 mg twice a day at Day 8, to 250 mg three times a day at Day 15, subject to reports of poor tolerance of gastrointestinal symptoms or other side effects.
  Arms: Lifestyle Intervention and Metformin
Behavioral: Intensive Lifestyle Intervention — The intensive lifestyle interventions for the Active Intervention groups will be done at the Lifestyle Intervention Centres. The aim would to achieve and maintain a weight reduction of at least 7 percent of initial body weight through a healthy reduced-calorie, low-fat diet and engagement in physical activity of moderate intensity for at least 150 minutes per week.
  This will be accomplished through a programme of individualized fitness assessment and exercise prescription for cardiovascular, strength and functional training that is standardized across study sites and facilities. The programme comprises an initial 32 sessions (2 times weekly) for supervised gym workout over 16 weeks, followed by maintenance programme of regular unsupervised exercises.
  Arms: Lifestyle Intervention and Metformin
Behavioral: Standard LIfestyle Recommendation — The standard lifestyle recommendations for the Control groups are in the form of standard diabetic education pamphlets and a 20-to-30-minute individual session that emphasizes the importance of a healthy lifestyle to reduce their weight and to increase their physical activity. Activity will be monitored using a pedometer.
  Arms: Standard Level of Care

SUMMARY:
Dementia (Alzheimer's Disease) is sometimes called "Type 3 Diabetes" because of the strong connection between Type 2 diabetes (a function of insulin resistance) with Dementia.

The investigators therefore hypothesize that Reducing Insulin Resistance using Intensive Lifestyle Intervention (Exercise and Weight loss) + Metformin Treatment in Prediabetic & diet-control-only Diabetic overweight and mildly cognitively impaired individuals 55 years or older would lead to better Cognitive Function (compared to standard care) after 2 years.

Subjects will be monitored and assessed using a battery of Cognitive and psychological tests and PET scans to demonstrate glucose utilization in the relevant areas of the brain.

This 3-year open-label study aims to recruit 360 subjects with 50% (180 subjects) randomized to receiving Intensive lifestyle intervention with Metformin (if diabetic) vs the other 50% who would receive only the usual standard level of care in the primary care setting.

DETAILED DESCRIPTION:
General Introduction In this trial, the drug to be studied is Metformin. It is an insulin-sensitizing biguanide which has long been used safely as an effective antidiabetic drug for patients with type II diabetes.

Rationale for the Study Purpose Dementia is a clinical syndrome due to multiple aetiologies, of which Alzheimer disease (AD) and Vascular Dementia (VaD) are the two most common. Dementia represents the advanced stage of a syndrome spectrum of cognitive impairment, an age-associated neurodegenerative condition that includes ageing related cognitive disorder (aka age-associated memory impairment or subject memory impairment, i.e. memory loss without other cognitive problems and are within normal limits given the person's age), and Mild Cognitive Impairment (MCI), a clinical entity that includes memory and cognitive impairment but no significant functional disability to meet threshold criteria for diagnosis of dementia. Of note, MCI is considered a prodromal state of dementia that increases the risk of subsequently developing dementia.

MCI can be classified into two main categories: (1) amnestic MCI and (2) non-amnestic MCI. Each MCI subtype can be further classified according to the presumed aetiology: degenerative; vascular; psychiatric; or traumatic.

1. Amnestic MCI (aMCI, prominent memory impairment with possibly mild degrees of impairment in other cognitive domains),
2. Non-amnestic MCI (non-aMCI, in which memory is largely unaffected but other domains of cognitive and behavioural functioning are impaired).

Currently available drugs approved for AD (anticholinesterases and Memantine) have limited efficacy and do not alter the pathophysiological basis of disease nor disease progression. No drugs are currently approved by regulatory authorities specifically for the treatment of MCI. Because treatments are less effective when the disease is far advanced, individuals with MCI at earlier stages of their illness are likely better candidates for clinical trials. Neuropathology-based studies of "clinically non-demented" individuals show high burdens of vascular and AD types of pathology. MCI may therefore be a pathologically-based preclinical or early clinical phase of dementia that is likely to progress to AD or VaD, and is hence an appropriate predementia syndrome for therapeutic intervention.

Vascular-related Risk Factors. Prior research up to date amply supports the hugely important role of vascular-related risk factors in the aetiology of both AD and VaD. Because vascular-related risk factors are treatable, it should be possible to prevent, postpone or mitigate VaD as well as AD (to the extent due to the vascular contribution of its aetiology). The vascular and related factors that have been associated with dementia and cognitive decline include diabetes and insulin resistance, high blood pressure (BP) and hypertension, total cholesterol and other lipid parameters, body mass index (BMI) and obesity, and the metabolic syndrome (MetS). MetS is a clustering of cardiovascular risk factors related to central obesity including impaired glucose metabolism, dyslipidaemia, and high BP that is associated with increased risk for both Type 2 Diabetes Mellitus (T2DM) and coronary artery disease (CAD). MetS has been shown to be associated with an increased risk of predementia syndromes including age-related cognitive decline, MCI and VaD, albeit with mixed findings of associations with AD. Insulin resistance is widely considered to play the central role in the pathophysiological mechanism of MetS. Hence, lifestyle and therapeutic interventions targeted at lowering insulin resistance is a promising MCI treatment option with the aim to slow cognitive decline and prevent or delay progression to dementia due to AD and/or VaD).

The role of insulin resistance in MCI and dementia Insulin and insulin resistance play important roles and functions in the central nervous system and the development of age-related neurodegenerative diseases, including glucose metabolism, vascular function, synaptic maintenance, beta-amyloid regulation, and tau phosphorylation. Insulin is transported across the blood-brain barrier, and brain insulin receptors are selectively localized in key brain regions, such as hippocampus, entorhinal cortex, and frontal cortex, where it plays a direct role in modulating levels of important neurotransmitters, synaptic plasticity, learning and memory. Insulin has also been shown to regulate the metabolism of beta-amyloid and tau, the building blocks of amyloid plaques and neurofibrillary tangles which are the neuropathological hallmarks of AD. Peripheral hyperinsulinemia promotes oxidative stress, protein glycosylation and cerebral ischemia and impairs the clearance of amyloid beta in the brain through competition for insulin degrading enzyme (IDE).

Diabetic patients are more likely to manifest impaired cognitive function, cognitive decline and a significantly higher risk of developing Alzheimer's disease or vascular dementia. Both hyperglycaemia and insulin resistance (IR) have also been shown in population-based studies to be associated with poor cognitive function in older persons. Hippocampal volumes were smaller in diabetic patients and in those with increased insulin resistance than in normal healthy controls. Several mechanisms are likely to explain the increased risk of cognitive impairment in T2D. Insulin resistance as mentioned above has been shown to play a direct role in cognitive impairment in individuals with type 2 diabetes (T2D). Additionally, chronic hyperglycaemia has been shown to be associated with decreased cerebral blood flow, decreased glucose transport across the blood brain barrier, reduced cerebral glucose metabolism and microvascular changes from endothelial damage. Finally, metabolic and vascular risk factors such as dyslipidaemia and hypertension which are closely linked to IR and T2D have been shown to predict cerebrovascular disease, cognitive decline and dementia.

Lowering Insulin Resistance Recent data support the development of therapeutics that target insulin pathways and particularly the lowering of insulin resistance as potential treatments for AD. Insulin administration reduces neuronal accumulation of beta-amyloid peptides and synaptic binding of toxic beta-amyloid derived diffusible ligands in cell culture; it improves cognitive performance in rodents and reportedly in patients with early AD. Insulin-sensitizers like peroxisome proliferator-activated receptor-gamma (PPAR- gamma) have been reported to improve insulin sensitivity, decrease inflammation and inhibit A-beta-stimulated secretion of pro-inflammatory products.

Rosiglitazone is a thiazolidinedione that stimulate PPAR-gamma and has been shown to inhibit beta-amyloid production. This insulin sensitizer is used as an oral drug (Avandia) effective in the treatment and prevention of diabetes. However, recent concerns about increased cardiovascular mortality has restricted its use in diabetic patients.

Initial reports suggest that Rosiglitazone is a promising drug in the treatment of AD. Positive effects on cognitive function have been reported in preclinical animal studies and a handful of preliminary clinical studies. However, these findings have not been confirmed subsequently by Phase III trials of patients with mild to moderate AD.

A growing consensus about treatment trials of AD is that they may be conducted at too late in the disease process for them to be effective.

Nevertheless an abundance of data strongly supports the central role of underlying metabolic pathogenesis in AD and VaD. Agents which modify insulin sensitivity remain as therapeutic options highly worthy of further inquiry. As rosiglitazone is a substrate for the multidrug-resistant gene product permeability glycoprotein, it may not have high penetration through the blood-brain barrier.

Metformin, however, is an insulin-sensitizing biguanide has long been used safely as an effective antidiabetic drug for patients with T2D and is the only antidiabetic drug that has been conclusively shown to prevent cardiovascular complications of diabetes. It has been shown that metformin evidently crosses the blood-brain barrier, accumulates in the brain and acts directly on the central nervous system.

A major mechanism of metformin action is activation of AMP-activated protein kinase (AMPK), which plays a key role in cellular energy homeostasis, insulin signalling, and the metabolism of glucose and fats. The activation of AMP-activated protein kinase and anti-inflammatory actions of metformin has been shown to occur not only in peripheral tissues but also in the brain.

There is hitherto no published report of the effect of metformin treatment on cognitive outcomes in diabetic patients. Recently, the investigators have completed a 4 year follow-up study of older diabetic patients and have found that long term metformin use of ≥6 years was prospectively associated with lower risk of cognitive impairment.

Metformin is an oral antidiabetic drug in the biguanide class. It is the first-line drug of choice for the treatment of type 2 diabetes, in particular, in overweight and obese people.

In this trial, the dosage schedule of metformin is only 250 mg thrice a day, (up-titrated weekly from a starting dose of 250 mg once a day). Despite its well-documented tolerability, this proposed weekly incremental dosage is designed to further reduce possible side-effects to drug-naive diabetic subjects taking Metformin for the 1st time.

Hypothesis The novel strategy of lowering insulin resistance with dietary modification and exercise in combination with a commonly used safe anti-diabetic medication, metformin could help to slow down cognitive decline and dementia.

Study Population Chinese patients are used as this proposed clinical trial builds upon and also uses the patients of our on-going Singapore Longitudinal Ageing Studies (SLAS) Study, where only Chinese Patients are used.

360 Chinese patients with prediabetes or diabetes with MCI will be identified and recruited from the community and primary care clinics in:

1. Singapore Longitudinal Ageing Studies (SLAS): SLAS-1 cohort in South East Region and SLAS-2 cohort in South West Region.
2. Marine Parade Polyclinic and Geylang Polyclinic.

Study Design Summary 24-month randomized controlled parallel-group study (IRMCI Study) of overweight-or-obese pre-diabetes older patients (IRMCI-1) or untreated type 2 diabetes (IRMCI-2) older patients, all with amnestic MCI or non-amnestic multi-domain MCI, will be randomly assigned within Apolipoprotein E4 (ApoE4) positive and ApoE4 negative strata to:

1. IRMCI-1 (prediabetic patients): Active Intervention (Intensive lifestyle modification) or Control group (standard lifestyle recommendations).
2. IRMCI-2 (diabetic patients): Active Intervention (Intensive lifestyle modification) plus metformin (Glucophage, 250mg thrice daily) or Control group (standard lifestyle recommendations).

Cognitive screening and diagnostic assessments are performed using the Mini mental State Examination (MMSE) and Montreal Cognitive Assessment scale (MoCA), and a comprehensive Neuropsychological Test Battery that will assess performance on multiple cognitive domains (Memory, Story Memory, Language, Executive function, Visual-Spatial and Constructional ability and Attention.)

The Subjects with age-and education-adjusted MMSE<26 or MOCA<26 or memory and non-memory domains test score that is 1.0 Standard Deviation (SD) or more below age-education adjusted norms are evaluated by Clinical Dementia Rating (CDR) scale. Subjects with a CDR global score of 0.5 together with Sum of Boxes of ≥3 or global score of ≥1 denoting dementia undergo a structured clinical assessment including neurologic examination, laboratory tests and final review by an expert panel of neurologists and psychiatrists, for final diagnosis and sub-classification of MCI, according to an standard SLAS protocol already established for the assessment and diagnosis of MCI and dementia.

Randomization:Subjects will be split into 2 Groups namely (1) Pre-Diabetic and (2) Diabetic. Each of these 2 groups will be stratified with APOE 4 allele as a stratification factor. .

The Prediabetic group will thus be similarly stratified into (B) Prediabetic-APOE4+ and (A) Prediabetic-APOE4-.

The Diabetic group will thus be stratified into (D) Diabetic-APOE4+ and (C) Diabetic-APOE4-.

Each of these four groups (A), (B), (C), & (D) will have their individual list of 360 randomization numbers generated by NUS Research Fellow using SAS computer programme. Each of these 360 x 4 numbers will be individually sealed in envelopes that will be numbered and used serially (from 0001st to 0360th for each group).

Subjects will have their Diabetic/Prediabetic status and APOE4+or- status determined using existing and baseline laboratory tests. They will then be assigned accordingly to the appropriate group [ ie (A), (B), (C), & (D)]. Trained nurses will then assign subjects to treatment vs control arm using the treatment allocation determined within the serially allotted sealed envelopes. .

There will not be any blinding as this is an open-labelled randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Singapore Citizen or Permanent Resident.
2. BMI of 23 or higher (Asian criteria for overweight and obese, Ministry of Health Recommendation, Singapore); and/or Waist Circumference: ≥ 90cm and ≥ 80cm for Chinese men and women respectively.
3. Prediabetes (if Not diabetic):

   * Impaired fasting glucose (IFG): (ADA criteria: fasting plasma glucose level from 5.6 mmol/L (100 mg/dL) to 6.9 mmol/L (125 mg/dL), and/or
   * Impaired glucose tolerance (IGT) (WHO and ADA criteria: two-hour glucose levels of 140 to 199 mg per dL (7.8 to 11.0 mmol) on the 75-g oral glucose tolerance test,. and/or
   * HbA1C: 5.7- 6.4% (ADA criteria)
4. Type 2 Diabetes (if Not prediabetic) yet to be treated with anti-diabetic drug treatment ('on diet control only'), with HbA1c <8.0% OR Diabetics who have been taken off medication for =/> 1 year with HbA1c< 8.0% will be considered for recruitment.

   * If HbA1c is 8.0- 8.4% at any follow-up visit, then try diet and lifestyle control and repeat at next visit (i.e. 3 months later). If 2 consecutive repeat HbA1c readings are still 8.0-8.4% or if subjects choose to start on or increase medication for diabetes, then take out of study and start medication.
   * If HbA1c =/>8.5% at any time after Recruitment, take out of study and start medication.
5. Mild Cognitive Impairment:

   * The individual is neither normal nor demented;
   * There is evidence of cognitive deterioration, shown by either objectively measured decline over time or subjective report of decline by self or informant in conjunction with objective cognitive deficits; and
   * Activities of daily life are preserved and complex instrumental functions are either intact or minimally impaired.
   * This will be operationalized in the study as:

     * A Subjective memory or cognitive complaint by the patient and/or by the caregiver
     * Objective cognitive deficit documented by performance on a battery of multiple-domain neuropsychological tests (See below): a score that is 1.0 SD or more below age- and education-adjusted local norms
   * aMCI: Deficit in delayed recall subtest of the Rey Auditory Verbal Learning Test (RAVLT) and Story Memory test
   * mdMCI: Deficit in language, executive function, visuospatial/constructional ability, block design, and attention.
   * Generally intact Activities of Daily Living as measured by Instrumental and Basic Activities of Daily Living (IADL and BADL).
   * No dementia:

Exclusion Criteria:

1. Contraindications to Metformin treatment: Creatinine of > 150umol/L, history of decompensated liver disease, liver cirrhosis, or unexplained elevated hepatic transaminases (ALT or AST >3x Upper Limit of Normal; Upper Limits as accepted by SingHealth Polyclinics as 66 U/L for ALT and 42 U/L). This contraindication would not affect Subjects with a history of high baseline ALT and/or AST which have been evaluated by a Hepatologist to be due to Non-alcoholic Fatty Liver Disease without cirrhosis.,
2. Severe Neuro-Musculoskeletal and Sensory Disabilities
3. Severe Psychiatric disorders (eg; alcohol abuse, severe depression, schizophrenia, bipolar disorder)
4. Illnesses that seriously reduce life expectancy or ability to participate in the trial
5. Congestive heart failure (New York Heart Association cardiac status classes 2, 3 or 4), Myocardial infarction or Coronary artery Bypass surgery or percutaneous coronary intervention within the past 6 months, Cardiac Arrhythmias, Severe Hypertension.
6. Concurrent use or recent use (within 1 week or 5 half lives of the drug whichever is longer) of drugs with anticholinesterase, sedating or central nervous system (CNS) side effects: antispasmodics, antiemetics, antidiarrhoeals, antihistamines, hypnotics, antidepressants, antipsychotics, bronchodilators.
7. Concurrent use of drugs (for >4 consecutive weeks) or use of drugs within 12 weeks of screening) that are known to adversely affect glucose tolerance and its interpretation: .
8. History of Hypersensitivity to any of the Study Drug or to Drugs of similar chemical classes
9. Use of an Investigative Drug within 30 days or 5 half-lives of the drug whichever is longer
10. Potentially Unreliable and/or judged by the investigator to be Unsuitable for the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint (Cerebral Glucose Metabolic Rate) | 2 years
  Change in Cerebral glucose metabolic rate & MRI Measures of Cerebral Volumetric and functional changes and white matter structural and functional connectivity as measured by Fluorodeoxyglucose Positron Emission Tomography & 3T MRI (FDG-PET/MRI) scans at Baseline and at 2 years.
Primary cognitive endpoint (Neuropsychological Performance) | 2 years
  Change in Composite z-score of memory and multi-domain non-amnestic cognitive test performance using a Neuropsychological Assessment performed at Baseline and at 2 years.

SECONDARY OUTCOMES:
Secondary clinical endpoints Subjective Memory and Cognitive Complaint (SMCC | 2 years
  Change in Subjective Memory and Cognitive Complaint (SMCC) as measured at baseline and at 2 years.
Secondary clinical endpoints Basic Activities of Daily Liver (ADL) | 2 years
  Change in Basic Activities of Daily Liver (ADL) as measured at baseline and at 2 years.
Secondary clinical endpoints Cognitive Instrumental Activities of Daily Living Scale | 2 years
  Change in Cognitive Instrumental Activities of Daily Living Scale (Cog-IADL) as measured at baseline and at 2 years.
Secondary clinical endpoints Global Clinical Dementia Rating Sum of Boxes | 2 years
  Change in Global Clinical Dementia Rating Sum of Boxes (version with Informant and version without need for Informant- CDR-SB) as measured at baseline and at 2 years.
Secondary clinical endpoints Mini-Mental State Examination | 2 years
  Change in Mini-Mental State Examination [MMSE]as measured at baseline and at 2 years.
Secondary clinical endpoints Montreal Cognitive Assessment scale | 2 years
  Change in Montreal Cognitive Assessment scale [MoCA] as measured at baseline and at 2 years.
Secondary adherence endpoints fasting plasma insulin | 2 years
  Markers of lowered insulin resistance (Change in fasting plasma insulin) as measured at baseline and at 2 years.
Secondary adherence endpoints Homeostatic Model Assessment (HOMA) | 2 years
  Markers of lowered insulin resistance [Change in Homeostatic Model Assessment (HOMA)] as measured at baseline and at 2 years.
Secondary adherence endpoints Lifestyle Intervention (Change in Weight) | 2 years
  Lifestyle Intervention (Change in Weight) as measured at baseline and at 2 years.
Secondary adherence endpoints Body Mass Index | 2 years
  Lifestyle Intervention [Change in Body Mass Index (BMI)] as measured at baseline and at 2 years.
Secondary adherence endpoints Waist Circumference | 2 years
  Lifestyle Intervention (Change in Waist Circumference) as measured at baseline and at 2 years.
Secondary adherence endpoints Fasting plasma glucose | 2 years
  Glycemic Control (Change in Fasting plasma glucose) as measured at baseline and at 2 years.
Secondary adherence endpoints Glycated Hemoglobin (HbA1c) | 2 years
  Glycemic Control [Change in Glycated Hemoglobin (HbA1c)] as measured at baseline and at 2 years.
Secondary adherence endpoints Fasting Lipids | 2 years
  Metabolic control [Change in Fasting Lipids (total cholesterol, HDL-Chol, LDL-Chol, triglycerides)] as measured at baseline and at 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: NG TZE PIN, MD, Principal Investigator — National University of Singapore
Locations (1):
- SingHealth Polyclinics - Marine Parade Polyclinic, Singapore, Singapore

REFERENCES:
- [Background] Pathan AR, Gaikwad AB, Viswanad B, Ramarao P. Rosiglitazone attenuates the cognitive deficits induced by high fat diet feeding in rats. Eur J Pharmacol. 2008 Jul 28;589(1-3):176-9. doi: 10.1016/j.ejphar.2008.06.016. Epub 2008 Jun 7. PMID 18602098
- [Background] Watson GS, Cholerton BA, Reger MA, Baker LD, Plymate SR, Asthana S, Fishel MA, Kulstad JJ, Green PS, Cook DG, Kahn SE, Keeling ML, Craft S. Preserved cognition in patients with early Alzheimer disease and amnestic mild cognitive impairment during treatment with rosiglitazone: a preliminary study. Am J Geriatr Psychiatry. 2005 Nov;13(11):950-8. doi: 10.1176/appi.ajgp.13.11.950. PMID 16286438
- [Background] Risner ME, Saunders AM, Altman JF, Ormandy GC, Craft S, Foley IM, Zvartau-Hind ME, Hosford DA, Roses AD; Rosiglitazone in Alzheimer's Disease Study Group. Efficacy of rosiglitazone in a genetically defined population with mild-to-moderate Alzheimer's disease. Pharmacogenomics J. 2006 Jul-Aug;6(4):246-54. doi: 10.1038/sj.tpj.6500369. Epub 2006 Jan 31. PMID 16446752
- [Background] Abbatecola AM, Lattanzio F, Molinari AM, Cioffi M, Mansi L, Rambaldi P, DiCioccio L, Cacciapuoti F, Canonico R, Paolisso G. Rosiglitazone and cognitive stability in older individuals with type 2 diabetes and mild cognitive impairment. Diabetes Care. 2010 Aug;33(8):1706-11. doi: 10.2337/dc09-2030. Epub 2010 Apr 30. PMID 20435794
- [Background] Gold M, Alderton C, Zvartau-Hind M, Egginton S, Saunders AM, Irizarry M, Craft S, Landreth G, Linnamagi U, Sawchak S. Rosiglitazone monotherapy in mild-to-moderate Alzheimer's disease: results from a randomized, double-blind, placebo-controlled phase III study. Dement Geriatr Cogn Disord. 2010;30(2):131-46. doi: 10.1159/000318845. Epub 2010 Aug 21. PMID 20733306
- [Background] Harrington C, Sawchak S, Chiang C, Davies J, Donovan C, Saunders AM, Irizarry M, Jeter B, Zvartau-Hind M, van Dyck CH, Gold M. Rosiglitazone does not improve cognition or global function when used as adjunctive therapy to AChE inhibitors in mild-to-moderate Alzheimer's disease: two phase 3 studies. Curr Alzheimer Res. 2011 Aug;8(5):592-606. doi: 10.2174/156720511796391935. PMID 21592048
- [Background] Ng TP, Feng L, Yap KB, Lee TS, Tan CH, Winblad B. Long-term metformin usage and cognitive function among older adults with diabetes. J Alzheimers Dis. 2014;41(1):61-8. doi: 10.3233/JAD-131901. PMID 24577463
- [Background] Brackett CC. Clarifying metformin's role and risks in liver dysfunction. J Am Pharm Assoc (2003). 2010 May-Jun;50(3):407-10. doi: 10.1331/JAPhA.2010.08090. PMID 20452916
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] American Diabetes Association. (6) Glycemic targets. Diabetes Care. 2015 Jan;38 Suppl:S33-40. doi: 10.2337/dc15-S009. No abstract available. PMID 25537705
- [Background] Standards of medical care in diabetes--2015: summary of revisions. Diabetes Care. 2015 Jan;38 Suppl:S4. doi: 10.2337/dc15-S003. No abstract available. PMID 25537706